CLINICAL TRIAL: NCT04746898
Title: Effectiveness Of Different Simulation Methods As A Training Strategy In Basic Life Support In Increasing Knowledge And Skills: A Randomised Control Trial
Brief Title: Effectiveness Of Different Simulation Methods As A Training Strategy In Basic Life Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Nurten Taşdemir Assoc. Prof. PhD. (Unknown)
Responsible Party: Principal Investigator, Dilek YILDIRIM TANK, Research Assistant, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZonguldakBEU
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Nurse's Role; Simulation Training; Cardiopulmonary Resuscitation
Keywords: Nurse; Simulation Training; Virtual Reality; High Fidelity Simulation; Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Training Group (VR group) (Experimental): The students in the first group received basic life support practice training with virtual reality applications.
  Interventions: Other: Virtual Reality Training
- High Fidelity Simulation Training Group (HFS group) (Experimental): The students in the second group received basic life support practice training with high fidelity simulators.
  Interventions: Other: High Fidelity Simulation Training
- Low Fidelity Simulation Training Group (LFS group) (Experimental): The students in the third group received basic life support practice training with the classical method, low-reality mannequin.
  Interventions: Other: Low Fidelity Simulation Training

INTERVENTIONS:
Other: Virtual Reality Training — Students received their basic life support application training through virtual reality glasses with special software.
  Other Names: High Fidelity Simulation Training
  Arms: Virtual Reality Training Group (VR group)
Other: High Fidelity Simulation Training — Students received their basic life support application training through high fidelity simulator mannequins.
  Arms: High Fidelity Simulation Training Group (HFS group)
Other: Low Fidelity Simulation Training — Students received their basic life support application training through low fidelity simulator mannequins.
  Other Names: Traditional Method
  Arms: Low Fidelity Simulation Training Group (LFS group)

SUMMARY:
The experimentally planned research was carried out with the students of Zonguldak Bülent Ecevit University Faculty of Health Sciences Nursing Department between 21.02.2020-02.09.2020.After the informed consent form was obtained from the students who accepted to participate in the study, the students were divided into three groups by applying block randomization with the computer-assisted randomization method. Then, all students filled in the Participant Identification Form and the Basic Life Support Application Steps for Adults Information Form. Later, with a visual-based presentation prepared in line with the guideline updated and published by the American Heart Association (AHA) in 2015, a 30-minute training on basic life support for adults was given.At the end of the training, the students were informed about the groups they were in, and the working principles of the devices the groups would work on were informed. With the first group virtual reality applied scenario, the 2nd group computer-aided scenario-based high-reality simulation device (SimMan® 3G) and the 3rd group low-reality adult basic life support model.The groups will be taken to the laboratories individually and the applications will be done individually and other students were not allowed to follow the student who did the application during the application. During the application, the students were evaluated with the basic life support application evaluation form. During the application, the video recording taken with the permission of the students was watched with the student after the application and a debriefing session was held. After the application, education was evaluated with Student Satisfaction and Self-Confidence in Learning Scale. Basic life support knowledge level was evaluated by having the basic life support information assessment form filled out again at 3 and 6 months after the first evaluation.

DETAILED DESCRIPTION:
Cardiac arrest is an important health problem and cause death all over the world. In the event of an arrest, the initiation of emergency resuscitation increases survival rates by 3-fold. Although basic life support is vital, unfortunately the level of knowledge on the subject is quite low. When the nursing programs are examined, it is seen that the first aid emergency care course is included in the nursing undergraduate education plan of Higher Education Institutions Core Program. It is seen that theoretical and clinical applications are carried out in the scope of First Aid and Emergency Care Nursing course.

Clinical practice is an essential part of nursing education. However, during clinical practice, factors such as inadequacy of clinical application areas, not feeling ready for students, fear of harming the patient and making mistakes, increasing student / instructor ratio increase the anxiety levels of students and thus prevent students from making patient care correctly and completely. During clinical practice, students should realize their practices by paying attention to the values and rights of the patients and it is very important to ensure patient safety.

Technological advances, which allow for the recurrence of clinical skills and the opportunity to experience rare clinical conditions, enable students to work with models that act as real patients in environments similar to actual clinical settings. While providing this, it is a teaching method that maintains the safety of the patient, improves the ability of skill by learning and provides learning opportunity without fear of harm to the patient. However, there are many positive features such as increasing students' motivation, encouraging learning and increasing self-confidence. Computer-aided simulation and virtual reality applications developed within the scope of experience-based teaching design are enriched with feedback and increase learning outcomes. Considering all these, the use of simulation practices and tools in nursing education is rapidly increasing.

The didactic teaching and learned procedures, which are among the various advantages of simulations, are considered as a learning tool that will increase the success in healthcare practices, thanks to the opportunity to apply them to patients. However, expensive simulators that are dependent on teaching in terms of design, space and feedback have accessibility problems. For this reason, this study has been planned in order to determine the method required to ensure effective education of vital first aid applications and firstly the basic life support application and to determine the most effective method to ensure the best integration into education in this rapidly advancing period of technology.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate the study,
* Having taken basic nursing education courses,
* Passing the Basic Principles and Practices in Nursing Course with a letter grade of CB and above
* Having taken basic English courses,
* Not having received first aid training before,
* To be able to speak and understand the Turkish language,
* Ability to use technological devices

Exclusion Criteria:

* Not wanting to participate in the study,
* Not taking basic nursing education courses,
* Getting CC and under letter grade from Basic Principles and Practices in Nursing course
* Not taking basic English lessons,
* Having received first aid training before,
* Inability to speak and understand Turkish language adequately,
* Inability to use technological devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-02-18 (Estimated)

PRIMARY OUTCOMES:
Decreasing mortality and morbidity rates by increasing knowledge and skills of basic life support. | 6 months
  Unfortunately, the level of knowledge of health professionals about the essential life support application is very low. Nursing students who are highly likely to encounter patients with basic life support indications due to their professions will have a positive effect on survival rates if they graduate competently on this subject.
To determine the most effective method by evaluating students' knowledge level on the subject with the basic life support information assessment form | 6 months
  Technological developments that allow the repetition of clinical skills and the opportunity to experience rare clinical situations offer students the opportunity to work with models that behave like real patients in environments similar to real clinical settings. Determining the effective method in the education of a practice that is of vital importance such as basic life support will contribute to the effective increase of knowledge and skills of healthcare professionals and students studying in this field. The knowledge level of students about basic life support will be evaluated with a knowledge assessment form.
Determining an effective education method by evaluating basic life support practice skills after the education of students with different simulation methods. | 6 months
  The basic life support training of the students was applied with different simulation methods. After the training, the basic life support practice skills of the students were evaluated with the practice evaluation form prepared according to the AHA 2015 guide. Determining the effective method will contribute to the effective acquisition of practical skills to students.
To increase students' self-confidence and satisfaction levels about the practice after basic life support practice training | 6 months
  The students of our age, known as the generation Z, grow up with technology. The integration of different technological developments into education attracts their attention and increases their motivation. This increases students' self-confidence and satisfaction levels after training. Increasing satisfaction and self-confidence increases students' interest in education and their learning capacity. Thus, the acquisition and permanence of information on the subject increases. Student Satisfaction and Self-Confidence Scale was used to measure students' levels of satisfaction and self-confidence. The highest score that can be obtained from the scale is 65 and the lowest score is 13. High score that can be obtained from the total of the scale indicates high satisfaction and self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months

REFERENCES:
- [Background] Aqel AA, Ahmad MM. High-fidelity simulation effects on CPR knowledge, skills, acquisition, and retention in nursing students. Worldviews Evid Based Nurs. 2014 Dec;11(6):394-400. doi: 10.1111/wvn.12063. Epub 2014 Sep 11. PMID 25213578